CLINICAL TRIAL: NCT01324791
Title: Laparoscopic Antireflux Surgery Versus Endoscopic Full-thickness Gastroplication for Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Public Hospital Zell am See (Other)
Other Study IDs: Zell02
Record Dates: First submitted 2011-03-26; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

ARMS (2):
- laparoscopic antireflux surgery (Active Comparator)
  Interventions: Procedure: anti-reflux surgery
- endoscopic full-thickness-gastroplication (Active Comparator)
  Interventions: Procedure: anti-reflux surgery

INTERVENTIONS:
Procedure: anti-reflux surgery

SUMMARY:
Endoscopic full thickness gastroplication (Plicator-Procedure) has the potential to be a safe and effective alternative to laparoscopic antireflux surgery (LARS)to improve symptoms of GERD. This prospective randomized study compares objective and subjective outcome parameters of Plicator with that of LARS.

ELIGIBILITY:
Inclusion Criteria:

* long history of GERD symptoms
* persistent or recurrent symptoms despite optimal medical treatment
* persistent or recurrent complications of GERD
* reduced quality of life owing to increasing esophageal exposure to gastric juice
* pathological values in the preoperative evaluated functional parameters.

Exclusion Criteria:

* any distinct hiatal hernia detectable by gastroscopy or barium radiography
* dysphagia
* esophageal strictures
* poor physical status (American Society of Anesthesiologists (ASA) scores III and IV) and pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- GPH Zell am See, Zell am See, Salzburg, Austria